CLINICAL TRIAL: NCT04201626
Title: Effectiveness of Adapted Enhanced Recovery After Surgery Protocol in Open Gynecologic Oncology Surgery: A Randomized Controlled Trial
Brief Title: Adapted ERAS in Gynecologic Oncology Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ERAS_GYNONC 01
Record Dates: First submitted 2019-12-03; First posted 2019-12-17 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Genital Neoplasm Malignant Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (Experimental)
  Interventions: Procedure: Adapted ERAS
- Control (No Intervention)

INTERVENTIONS:
Procedure: Adapted ERAS — Each woman in the intervention group will attend a preoperative counseling session with nurse and doctors. In addition to the standard preoperative counseling, explaining the purpose, process, and the importance of ERAS protocol compliance will be added to the session. Preoperative nutrition and laboratory assessment will be done according to adapted ERAS protocol on that same visit.
  During admission, the intervention group participants are provided with care according to adapted ERAS protocol including no bowel preparation, no extended fasting before surgery, balanced intravenous crystalloid, thromboprophylaxis, multimodal pain control reducing opioid usage, multimodal anti-emetics medications, stepping diet up to regular diet within 24 hours, chewing gum for post-operative ileus prevention, early removal of Foley's catheter, and promote early ambulation using care checklist plan.
  Arms: ERAS

SUMMARY:
Background: In recent decades, the new concept of Enhanced Recovery After Surgery (ERAS) program has been well accepted in the fields of gynecologic surgery. Many studies have shown the effectiveness of ERAS protocol in reducing hospital's length of stay, patient's morbidity, and rate of postoperative complications while cutting back on health care cost. Thus, standard guidelines such as ACOG has strongly recommended ERAS protocol implementation into each institution. However, institutions have self-limitations on adapting the standard ERAS pathway published from ERAS society due to the demand in resources. The concept of partial implementation of ERAS protocol has been raised and was mentioned in guidelines that ERAS implementation should be individualized to each institution. Nevertheless, the effectiveness of adapted ERAS protocol itself has not been well researched.

Objectives: To examine the effect of partial implementation of ERAS protocol adapted to our institution on patient's recovery (based on hospital length of stay, pain score, time to flatulence, postoperative complications, and re-visits) compared to standard routine care in women diagnosed with gynecologic malignancy (cervix, endometrium, and ovary) undergoing elective open surgery.

Design: A randomized controlled trial in gynecologic cancers (cervix, endometrium, and ovary) women, age 18-75 years, undergoing elective open gynecologic oncology surgery at Faculty of Medicine, Chiang Mai University hospital. The participants will be randomly assigned into one of two study groups: intervention (adapted ERAS protocol) and control (standard routine care).

For the intervention group, each woman will be brought through the adapted ERAS protocol step by step starting from preoperative counseling and preparation, intraoperative management, and postoperative management standard according to the adapted ERAS protocol. For the control group, each woman will be cared for using routine standard care.

The primary outcome is length of hospital stay.

1.3 Proposed duration 24 Months

ELIGIBILITY:
Inclusion Criteria:

* 18 - 75 years old
* Diagnosed with gynecologic malignancy of cervix, endometrium, or ovary
* Elective laparotomy surgery

Exclusion Criteria:

* Intraoperative accidental injury to urinary or GI organs
* Retain endotracheal intubation after surgery
* Peritoneal drainage for monitoring of bleeding/infection
* Unable to follow oral instructions
* Severe neuromuscular disease
* Preoperative hyperalimentation
* Neoadjuvant chemotherapy within 3 weeks prior to the procedure
* Previous abdominal/pelvic radiation
* Bowel obstruction
* Emergency operation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | Through hospital discharge, an average of 5 days
  Length of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, MSc, Principal Investigator — Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiewhatpong P, Charoenkwan K, Smithiseth K, Lapisatepun W, Lapisatepun P, Phimphilai M, Muangmool T, Cheewakriangkrai C, Suprasert P, Srisomboon J. Effectiveness of enhanced recovery after surgery protocol in open gynecologic oncology surgery: A randomized controlled trial. Int J Gynaecol Obstet. 2022 Nov;159(2):568-576. doi: 10.1002/ijgo.14211. Epub 2022 Apr 21. PMID 35396709